CLINICAL TRIAL: NCT05552235
Title: Assessment of the Safety and Performance of an Elbow Brace in the Prevention of Injuries During Sports Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Decathlon SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: elbowSOFT300
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Epicondylitis; Tendonitis Elbow; Elbow Injury
MeSH Terms: conditions — Elbow Injuries | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthosis group (Experimental): Use of Elbow Soft 300 device during sport practice
  Interventions: Device: Elbow SOFT 300
- Control group (Other): No medical device used during sport practice
  Interventions: Other: Control group

INTERVENTIONS:
Device: Elbow SOFT 300 — 15 patients will be included in this group and will used the medical device ElbowSOFT 300 during sport practice (at least 2 sport sessions per week), for 6 weeks.
  Arms: Orthosis group
Other: Control group — 15 patients will be included in this control group and will performed their sport sessions as usual (without the medical device), for at least 2 sport sessions per week during 6 weeks.
  Arms: Control group

SUMMARY:
Decathlon has developed the Elbow soft300 which is a medical device that must be positioned around the elbow to keep a physical activity on a regular basis in case of chronic epicondylitis, pain associated with tendonitis or chronic instability.

The objective of this multicentre study is to collect data on the related clinical complications and clinical outcomes of market-approved Decathlon Elbow soft 300 product to demonstrate safety and performance of this device in a real-world setting.

Outcome data collected from this study will provide the basis for Post-Market Surveillance (PMS) reporting, Clinical Study Report (CSR), Clinical Evaluation Report (CER) on Decathlon ElbowSoft300 device and support peer-reviewed publications on products performance and safety.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 18 years old
* Subject has a chronic epicondylitis (>3 months) OR elbow pain associated with tendonitis OR chronic elbow instability (>3 months)
* The current condition of his/her elbow allows the subject to continue usual physical activity
* Subject has been informed and is willing to sign an informed consent form
* Subject is willing to comply with protocol requirements and return to the study center for all clinical evaluations and required follow-up (6 weeks)
* Subject is affiliated to the French social security regime

Exclusion Criteria:

* Subject has conditions that may interfere with his/her ability to understand protocol requirements, participate in scheduled visits, or provide his/her informed consent
* Subject has worn a support (elbow brace or articulated orthosis) in the last month during his/her sport practice
* Subject has any medical condition that could impact the study at investigator's discretion
* Subject has a known hypersensitivity or allergy to the components of the device (polyamide, elastodiene, polyester, elastane)
* Adult subject to legal protection measure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Functionnal score | Change from Baseline functionnal score at 6 weeks
  Comparison of the Patient Rated Elbow Evaluation (20-item questionnaire with a global score from 0=best outcome to 100=worst outcome) between the baseline and last follow-up visit in each group (orthosis vs control)

SECONDARY OUTCOMES:
Confidence level (confidence questionnaire related to physical activity) | Change from Baseline confidence level at 6 weeks
  Gap in the confidence level related to physical activity (6-item questionnaire with a global score from 0=worst outcome to 100=best outcome), between the baseline and last follow-up visit in each group (orthosis vs control)
Elbow pain | Change from Baseline elbow pain at 6 weeks
  Comparison of elbow pain, assessed through a Numerical Rating Scale (NRS) ranging from 0=best outcome to 10=worst outcome, between the groups (orthosis vs control)
Elbow instability | Change from Baseline elbow instability at 6 weeks
  Comparison of elbow instability, assessed through a Numerical Rating Scale (NRS) ranging from 0=best outcome to 10=worst outcome, between the groups (orthosis vs control)
Safety (adverse events) | 6 weeks of follow-up
  Comparison of adverse events rates between the groups (orthosis vs control)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WIECZOREK, Principal Investigator — Centre Hospitalier Universitaire de Lille
Locations (2):
- France (2):
  - Centre Hospitalier de Boulogne-sur-Mer, Boulogne-sur-Mer
  - Centre Hospitalier Universitaire de Lille, Lille

IPD SHARING:
Plan to Share IPD: No